CLINICAL TRIAL: NCT00801268
Title: Randomized Clinical Trial of Triptolide Woldifii for Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: Randomized Clinical Trial of Triptolide Woldifii for Autosomal Dominant Polycystic Kidney Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: high rate of drop-out
Sponsor: Zhi-Hong Liu, M.D. (Other)
Responsible Party: Sponsor-Investigator, Zhi-Hong Liu, M.D., professor, Nanjing University School of Medicine
Organization: Nanjing University School of Medicine (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0802
Record Dates: First submitted 2008-11-25; First posted 2008-12-03 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Polycystic Kidney
Keywords: polycystic kidney disease; tripterygium wilfordii
MeSH Terms: conditions — Polycystic Kidney Diseases | interventions — Emodin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- emodin (Active Comparator)
  Interventions: Drug: Emodin
- Triptolide Woldifii (Experimental): TW60mg/d
  Interventions: Drug: tripterygium wilfordii

INTERVENTIONS:
Drug: tripterygium wilfordii — TW，60mg/d
  Arms: Triptolide Woldifii
Drug: Emodin — 100mg/d
  Other Names: Frangula emodin,Frangulic acid
  Arms: emodin

SUMMARY:
Triptolide has been approve effective in animal model.

DETAILED DESCRIPTION:
Randomized

ELIGIBILITY:
Inclusion Criteria:

* Clinically established ADPKD
* eGFR>30ml/min.
* Chinese nationality

Exclusion Criteria:

* Uncontrolled infections
* Non-ADPKD complications

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2008-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
MRI calculated kidney volume, eGFR | Every 3-6months

SECONDARY OUTCOMES:
End-stage kidney disease (ESRD) | every 2months

CONTACTS AND LOCATIONS:
Overall Officials: Liu Zhihong, Master, Principal Investigator — Research Institute of Nephrology, Jinling Hospital
Locations (2):
- China (2):
  - Liu ZH, Yao XD,Chen X,Hu YL, Nanjing, Jiangsu
  - Yao Xiaodan, Nanjing, Jiangsu